CLINICAL TRIAL: NCT04254289
Title: Pilot Randomized Trial of Ambulatory Exercise in Pulmonary Hypertension
Acronym: PaRTAkE-PH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Michigan (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Thomas Matthew Cascino, Clinical Lecturer in Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00150343
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Exercise; Six-minute walk; Heart rate monitor
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: An independent statistician will develop the randomization schedule and an unblinded study team member will document and maintain the treatment assignment log. The investigators will be adjusting the exercise regimens of those randomized to the exercise program and are unable to be blinded. All patients will receive weekly telephone calls to review activity logs. Outcomes included in the primary and secondary analysis will be blinded as possible. The staff performing the 6-minute walk test (6MWT) and interpreting echocardiograms will be blinded to the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual care administered at the Pulmonary Arterial Hypertension (PAH) clinic at the University of Michigan.
  Interventions: Behavioral: Usual Care
- Home-based exercise program (Experimental): Home-based individualized exercise program based on heart rate reserve (HRR).
  Interventions: Behavioral: Home-based exercise program

INTERVENTIONS:
Behavioral: Usual Care — Usual care
  Arms: Usual Care
Behavioral: Home-based exercise program — Home-based program determined by exercise physiologist
  Arms: Home-based exercise program

SUMMARY:
The researchers are investigating if changing an individual's behaviors may have an impact on outcomes for patients with pulmonary arterial hypertension (PAH). This research will test the efficacy of a home-based exercise program to improve exercise tolerance and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of group 1 Pulmonary Atrial Hypertension (PAH) diagnosed during right heart catheterization (RHC) according to WHO criteria 28
* WHO functional class II to III
* Stable clinical condition, with no change in medical therapy for pulmonary arterial hypertension (PAH) for at least 3 months before enrollment
* Planned follow-up at University of Michigan Hospital Centers over at least 1 year
* If enrolled in clinical trial, must be in open-label extension stage on stable medications for at least 3 months.
* Competent to give informed consent
* Have computer and internet access

Exclusion Criteria:

* Life expectancy under 1 year
* Co-morbidities which limit physical activity to a severe degree (i.e., permanently wheelchair bound, musculoskeletal disorders, recent myocardial infarction, unstable arrhythmia)
* Current substance abuse, and/or a severe psychiatric disorder (including severe depression, psychosis, or dementia) which limits the patient's ability to follow the study protocol
* Recently completed (<6 months), current enrollment or planned enrollment in pulmonary rehab.
* ≥30 minutes of exercise, ≥ 1 day per week for the previous 3 months
* Six-minute walk distance <150 meters or >550 meters
* Moderate or severe obstructive lung disease forced expiratory volume/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 65% of predicted value after bronchodilator administration).
* Moderate or severe restrictive lung disease (total lung capacity < 60% predicted value).
* Arterial oxygen saturation (SpO2) <88% during 6-minute walk test on baseline home oxygen prescription if applicable or SpO2 <80% if uncorrected shunt.
* History of exercise-induced syncope or arrhythmias.
* Pregnancy or lactation
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a home-based exercise training as measured by change in six-minute walk distance | Baseline, 12 weeks
  Distance measured in meters

SECONDARY OUTCOMES:
Efficacy of a home-based exercise training as measured by change in six-minute walk distance | Baseline, 6 months
  Distance measured in meters
Change in physical activity as measured by daily activity captured using the pedometer step count | Baseline, 12 weeks
  average daily step counts measured by a pedometer
Change in physical activity as measured by daily activity captured using the pedometer step count | Baseline, 6 months
  average daily step counts measured by a pedometer
Efficacy of a home-based exercise training as measured by change in treadmill exercise time | Baseline, 12 weeks
Efficacy of a home-based exercise training as measured by change in survey score from the EuroQol five dimension, five level (EQ-5D-5L) questionnaire. | Baseline, 12 weeks
  Health related quality of life assessed using the EuroQol EQ-5D-5L. There is a descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The survey visual analog scale (VAS) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
  The users guide gives details of the scoring system: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L_UserGuide_2015.pdf
Efficacy of a home-based exercise training as measured by change in survey score from the EuroQol five dimension, five level (EQ-5D-5L) questionnaire. | Baseline, 6 months
  Health related quality of life assessed using the EuroQol EQ-5D-5L. There is a descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The survey visual analog scale (VAS) records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
  The users guide gives details of the scoring system: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-5L_UserGuide_2015.pdf
Efficacy of a home-based exercise training as measured by change in survey score The Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) | Baseline, 12 weeks
  PAH-SYMPACT (Pulmonary Arterial Hypertension-Symptoms and Impact) is a self-rating questionnaire to assess symptoms and their physical and cognitive/emotional impact. The PAH-SYMPACT™ questionnaire consists of four domains: Cardiopulmonary Symptoms Domain (scored 0-24), Cardiovascular Symptoms Domain (scored 0-20), Physical Impacts Domain (scored 0-28), and the Cognitive/Emotional Impacts Domain (scored 0-16). In each domain a higher score indicates worse symptoms.
Efficacy of a home-based exercise training as measured by change in survey score The Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) | Baseline, 6 months
  PAH-SYMPACT (Pulmonary Arterial Hypertension-Symptoms and Impact) is a self-rating questionnaire to assess symptoms and their physical and cognitive/emotional impact. The PAH-SYMPACT™ questionnaire consists of four domains: Cardiopulmonary Symptoms Domain (scored 0-24), Cardiovascular Symptoms Domain (scored 0-20), Physical Impacts Domain (scored 0-28), and the Cognitive/Emotional Impacts Domain (scored 0-16). In each domain a higher score indicates worse symptoms.
Efficacy of a home-based exercise training as measured by change in survey score International Physical Activity Questionnaire Short Form (IPAQ-SF) | Baseline, 12 weeks
  The IPAQ-SF is 4 generic item questionnaire (7 questions). About physical activity time in the past 7 days.
Efficacy of a home-based exercise training as measured by change in survey score International Physical Activity Questionnaire Short Form (IPAQ-SF) | Baseline, 6 months
  The IPAQ-SF is 4 generic item questionnaire (7 questions). About physical activity time in the past 7 days.
Efficacy of a home-based exercise training as measured by change in survey score Patient Health Questionnaire (PHQ)-8 | Baseline, 12 weeks
  The PHQ-8 questionnaire about depression and is 8 items long. Each question ranges from 0 (not at all) to 3 (nearly every day) for a total possible score of 24 where higher score means more burdensome.
Efficacy of a home-based exercise training as measured by change in survey score Patient Health Questionnaire (PHQ)-8 | Baseline, 6 months
  The PHQ-8 questionnaire about depression and is 8 items long. Each question ranges from 0 (not at all) to 3 (nearly every day) for a total possible score of 24 where higher score means more burdensome.
Efficacy of a home-based exercise training as measured by change in World Health Organization (WHO) functional class | Baseline, 12 weeks
  The World Health Organization (WHO) functional class system was created to define the severity of an individual's symptoms and how they impact on day-to-day activities. The functional classes range from I to IV with IV having worse daily impairments.
Efficacy of a home-based exercise training as measured by change in World Health Organization (WHO) functional class | Baseline, 6 months
  The World Health Organization (WHO) functional class system was created to define the severity of an individual's symptoms and how they impact on day-to-day activities. The functional classes range from I to IV with IV having worse daily impairments.

OTHER OUTCOMES:
Change in heart rate recovery | Baseline, 12 weeks
Change in echocardiographic assessment of right ventricle size | Baseline, 12 weeks
Change in echocardiographic assessment of right ventricle function | Baseline, 12 weeks
Percent change in brain natriuretic peptide | Baseline, 12 weeks
Change in number of low risk criteria | Baseline, 12 weeks
  Criteria include: World Health Organization (WHO) functional class I/II, six-minute walk distance >440 m, brain natriuretic peptide (BNP) <50)
Frequency of completion of activity logs | Up to 12 weeks
Frequency of completion of weekly telephone follow-ups | Up to 12 weeks
Number of low risk criteria | 6 months
  Criteria include: World Health Organization (WHO) functional class I/II, six-minute walk distance >440 m, brain natriuretic peptide (BNP) <50
Number of hospitalizations for pulmonary hypertension | 12 weeks
Number of hospitalizations for pulmonary hypertension | 6 months
Frequency of Death | Up to 12 weeks
Frequency of Death | Up to 6 months
Frequency worsening WHO functional class | 12 weeks
  WHO functional class higher than previously noted. The World Health Organization (WHO) functional class system was created to define the severity of an individual's symptoms and how they impact on day-to-day activities. The functional classes range from I to IV with IV having worse daily impairments.
Frequency worsening World Health Organization (WHO) functional class | 6 months
  WHO functional class higher than previously noted. The WHO functional class system was created to define the severity of an individual's symptoms and how they impact on day-to-day activities. The functional classes range from I to IV with IV having worse daily impairments.
Frequency of need for escalation of pulmonary hypertension therapy | Up to 12 weeks
  Escalation implies dose increase is define as increase of existing therapy or addition of new medication for pulmonary arterial hypertension.
Frequency of need for escalation of pulmonary hypertension therapy | Up to 6 months
  Escalation implies dose increase is define as increase of existing therapy or addition of new medication for pulmonary arterial hypertension.
Frequency of syncope | 12 weeks
Frequency of syncope | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cascino, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No